CLINICAL TRIAL: NCT03546179
Title: Effect of Tidal Volume Challenge on Reliability of Plethysmography Variability Index in Hepatobiliary and Pancreatic Surgeries.
Brief Title: Tidal Volume Challenge and Reliability of Plethysmography Variability Index
Status: Completed | Type: Observational
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Hany M Yassin, MD, Associate professor, Fayoum University Hospital
Other Study IDs: D154
Record Dates: First submitted 2018-05-08; First posted 2018-06-06 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Abdominal Cancer
Keywords: PVI, Tidal volume challenge

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: tidal volume challenge test — Tidal volume (VT) will be increased from 6 to 8 ml/kg of for one minute and hemodynamic variables, including PVI with 8 ml/kg tidal volume ventilation (PVI8) will be recorded.
Other: Volume loading — After these two baseline hemodynamic measurements, volume expansion will be performed for 10 min using an infusion of balanced crystalloid solution (6ml/kg of predicted body weight).

SUMMARY:
The aim of this study is to investigate whether a temporary increase in tidal volume can predict fluid responsiveness in patients receiving a low tidal volume ventilation in hepatobiliary and pancreatic surgeries.

The hypothesis of this study is that a temporary increase in tidal volume from 6 to 8 ml/kg would improve the predictability of PVI in patients receiving low tidal volume ventilation in surgical procedures with large fluid shift as hepatobiliary and pancreatic procedures.

DETAILED DESCRIPTION:
Common hepatobiliary and pancreatic procedures include repair of lacerations, drainage of abscesses, and resection of primary or metastatic neoplasms. Care of patients undergoing hepatobiliary and pancreatic surgeries in the perioperative period is often challenging because of coexisting medical problems and debilitation found in many patients and because of the potential for significant operative blood loss. Hepatobiliary and pancreatic surgeries have been associated with high mortality and morbidity rates, but recent advances in anesthetic and surgical management have significantly reduced the operative risk.

Studies have shown that intraoperative optimization of cardiac output by repeated volume loading reduces postoperative morbidity and shortens hospital stay following abdominal surgery. However, unnecessary intravenous fluids may be deleterious, and intraoperative fluid restriction has been shown to improve clinical outcomes. During major hepatobiliary and pancreatic surgeries, intravascular volume expansion is constantly required but the safety margin of fluid management is quite narrow. The thought of fluid responsiveness has been progressively used in order to improve the fluid management of critically ill patients. Over the past two decades, many studies have been performed searching for the best index to predict fluid responder in a variety of clinical situations. recent studies have shown that what is called dynamic indexes of fluid responsiveness such as stroke volume variation (SVV), pulse pressure variation (PPV) and others are obviously superior to the more commonly measured static preload variables e.g. pulmonary artery occlusion pressure and central venous pressure.

Plethysmography variability index (PVI) is a dynamic variation parameter that automatically and continuously calculates the respiratory variations in the plethysmographic waveform acquired by the pulse oximeter. The PVI is presented as a safe and useful parameter for evaluating the fluid responsiveness of perioperative patients who underwent major abdominal surgery and for critically ill patients. Several studies have shown that PVI may predict fluid responsiveness in patients undergoing noncardiac surgeries as well as those under mechanical ventilation in the intensive care unit. However, the accuracy of the PVI is unclear for hepatobiliary and pancreatic operations that may have major cardiovascular changes and/or hyperdynamic circulation. Also, there are still limited studies investigating the direct relationship of PVI and cardiac preload status.

PVI is based on the respiratory variations in the pulse oximetry plethysmographic waveform amplitude and various factors that affect lung mechanics, including tidal volume (VT) could also influence PVI values and It is presumed that the effect of tidal volume reaches significance at >8 mL/kg Several studies have shown that dynamic indicators of fluid responsiveness do not reliably predict fluid response during low tidal volume ventilation whereas there is currently a growing trend towards a reduction in tidal volume, not only in ICU patients with acute lung injury but also in patients with healthy lungs undergoing surgery.

The 'tidal volume challenge' is a novel test proposed to improve the reliability of dynamic indexes in predicting fluid responsiveness in patients receiving low tidal volume ventilation. In a recent study testing the tidal volume challenge on some dynamic indexes, it is found that the changes obtained by transiently increasing tidal volume (tidal volume challenge) are superior to dynamic index itself in predicting ﬂuid responsiveness during low tidal volume ventilation. However, no studies use this novel test to know the reliability of PVI in predicting fluid responsiveness in patients receiving low tidal volume ventilation.

This study will be performed on adult patients undergoing hepatobiliary and pancreatic operations after obtaining approval of the Ethical and Scientific Committee of Fayoum University Hospital and National Liver Institute and written informed consent from the patients or their surrogates to participate. This study will be conducted at the National Liver Institute Hospital, Menoufia, Egypt.

Anesthetic technique:

On the day of surgery, intravenous access will be obtained. Demographic and anthropometric data will be recorded. All patients will be monitored by standard routine monitoring which includes a 5-lead electrocardiography, a non-invasive blood pressure, pulse oximetry, capnography, fractional inspired oxygen concentration (FiO2) and core temperature (using a nasopharyngeal probe). After preoxygenation, general anesthesia will be induced with Propofol 2 mg/kg IV, Fentanyl 1 µg/kg IV and Rocuronium 0.6 mg/kg IV followed by the endotracheal intubation. Maintenance of general anesthesia with a mixture of Sevoﬂurane with 50% oxygen in the air (GE Datex-Ohmeda S/5 Anesthetic Delivery Unit System). Mechanical ventilation will be performed in all patients on a semi-closed system adjusted to keep SaO2>95% and end-tidal CO2 between 35 mmHg and 40 mmHg.

A 7 F triple lumen central venous catheter will be inserted in the right internal jugular vein by ultrasound guidance. The central venous catheter will be connected to a pressure transducer, and the pressure trace will display continuously. The left radial artery will be cannulated, Pressure transducer will be placed on the midaxillary line and fixed to the operating table in order to keep the transducer at an atrial level during the study protocol. All transducers will be zeroed to atmospheric pressure for measuring invasive arterial blood pressure. An indwelling urinary bladder catheter will be inserted to monitor urinary output. Head and extremity wraps and warmer systems in the form of forced warming system (Model 750-Bair Hugger Temperature Management Unit, Arizant Healthcare Inc, USA) will be applied to maintain body temperature. A trans-esophageal Doppler (TED) probe (Cardio QP EDM™; Deltex Medical, Chichester, UK) will be greased with a lubricating gel and passed nasally into the mid-esophagus until aortic blood ﬂow signals will be best identified. Four skin electrodes (iSense electrical cardiometry skin sensors; Osypka Medical) will be applied on the neck and thorax per manufacturer recommendations on patients and electrical cardiometry monitor (electrical cardiometry monitor, ICON Cardiotronics, Inc., La Jolla, CA 92307; Osypka Medical GmbH, Berlin, Germany) will be connected to the sensor cable. These systems enable the continuous monitoring of stroke volume (SV), stroke volume Index (SVI), heart rate (HR), cardiac output (CO), cardiac index (CI), thoracic fluid content (TFC), systemic vascular resistance(SVR), corrected flow time (FTc) and stroke volume variation (SVV).

The Masimo Pulse Co-Oximeter probe (Masimo SET Rainbow R2-25r and R225a, Masimo Corp., Irvine, CA, USA) will be placed on the index finger of the patients and will be covered with a shield to eliminate light interference, as recommended by the manufacturer. The PVI and perfusion index (PI) variations will be automatically measured using the Masimo monitor (Masimo Radical-7, Masimo Corp., Irvine, CA, USA) with PVI software. PVI is an automatic measure of the dynamic change in PI that occurs during a complete respiratory cycle.

All throughout surgery packed red blood cells (300 ml) will be transfused when hematocrit percentage will be <25%. Fresh frozen plasma (unit of 200 ml) will be administrated when a Partial thromboplastin time>70 s, Fibrinogen <2 g/dl, or International Normalized Ratio (INR) >2. Patients will be extubated either in the operating room or post-operatively in intensive care unit.

Intervention protocol Initially, demographic data of patients including age, sex, height, actual body weight, predicted body weight (PBW), smoking history, comorbid diseases, operative time will be recorded.

After resection phase of tumours, baseline hemodynamic and respiratory variables including CI, CO, SV, SVI, SVV, SVR, HR, mean arterial pressure (MAP), central venous pressure (CVP), plateau pressure (Pplat), compliance of the respiratory system (Crs), TFC, FTc, PI and PVI with an 6 ml/kg tidal volume ventilation (PVI6) will be recorded. After baseline measurement, VT will be increased from 6 ml/kg to 8 ml/kg of predicted body weight for one minute and the above-mentioned hemodynamic variables, including PVI with 8 ml/kg tidal volume ventilation (PVI8) will be recorded. The tidal volume will be decreased back to 6 mL/kg PBW and after one minute measurements will be recorded. After these hemodynamic measurements, volume expansion will be performed for 10 min using an infusion of balanced crystalloid solution (6ml/kg of predicted body weight). The same hemodynamic parameters will be measured under ventilation with a VT of 6 ml/kg 5 min after volume loading. Thereafter the absolute (ΔPVI6-8,) and percentage change (%ΔPVI6-8) between the PVI at 6 mL/kg PBW (PVI6) and at 8 mL/kg PBW (PVI8) i.e. after performing a "tidal volume challenge" will be calculated. The change in PVI after giving the fluid bolus (ΔPVIfb) will also be calculated.

No more than two tidal volume challenges can be performed in any patient. Doses of vasoactive medications and PEEP will be kept constant.

STATISTICAL ANALYSIS:

Statistical analysis will be performed using SPSS version 24.0 (IBM, Armonk, NY, USA). Data are presented as mean (SD), median [interquartile range (IQR)], or number of patients (%). Changes in continuous variables from 6 to 8mL/kg PBW will be compared using paired t-test or Wilcoxon signed rank sum test, and group comparisons between responders and non-responders will be made using independent t-test or Mann-Whitney U test, as appropriate. Distribution normality will be assessed using the Shapiro-Wilk test. Categorical variables will be analyzed using chi-square test or Fisher exact test.To test the abilities of dynamic preload indices to predict fluid responsiveness, areas under the receiver operating characteristics (ROC) curves of the responders will be calculated and compared using the Hanley-McNeil test [area under the curve (AUC)=0.5, no better than chance, a useless test with no prediction possible; AUC=0.6-0.69, a test with a poor predictability; AUC=0.7-0.79, a fair test; AUC=0.8-0.89, a test with a good predictability; AUC=0.9-0.99, an excellent test; AUC=1.0, a perfect test with the best possible prediction]. A value of optimal threshold will be determined for each variable to maximize the Youden index [sensitivity + (specificity - 1)] For the sample size calculation, Statstodo computer program is used to calculate the sample size requirement for comparing two ROC curves with expected areas under the curves of 0.65 (PVI6) and 0.90 (ΔPVI6-8), assuming an α error of 0.05 and power of 90%, a minimum of 40 patients will be needed to detect an AUC difference of 0.25 when assuming the number of responders is similar to that of non-responders. The investigators expect data loss to be 20%, so 48 patients needed to be enrolled in this study

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years undergoing hepatic, pancreatic or biliary tumor resection

Exclusion Criteria:

* Preoperative cardiac arrhythmias
* Peripheral vascular disease
* Low left ventricular function (ejection fraction < 40%)
* Significant valvular heart disease
* Intra-cardiac shunts
* Pulmonary hypertension
* Fulminant hepatic failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years undergoing hepatic, pancreatic or biliary tumor resection
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
detection of best cut-off value of ΔPVI6-8 by using tidal volume challenge. | 2 minutes after performing a "tidal volume challenge"
  By Youden index [sensitivity + (specificity - 1)]

SECONDARY OUTCOMES:
Detection of sensitivity of PVI6 measured by masimo radical 7 equipment.. | 2 minutes before tidal volume challenge when tidal volume of patient is 6ml/kg
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of PVI6 measured by masimo radical 7 equipment.. | 1 minute before tidal volume challenge when tidal volume of patient is 6ml/kg
  By areas under the receiver operating characteristics (ROC) curves
Detection of best cut off of percentage ΔPVI6-8 measured by masimo radical 7 equipment. | 2 minutes after performing tidal volume challenge
  By areas under the receiver operating characteristics (ROC) curves and Youden index [sensitivity + (specificity - 1)]
Detection of sensitivity of ΔPVI6-8 measured by masimo radical 7 equipment. | 2 minutes after performing tidal volume challenge
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of percentage ΔPVI6-8 measured by masimo radical 7 equipment. | 2 minutes after performing tidal volume challenge
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of ΔPVI6-8 measured by masimo radical 7 equipment. | 2 minutes after performing tidal volume challenge
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of percentage ΔPVI6-8 measured by masimo radical 7 equipment. | 2 minutes after performing tidal volume challenge
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of PVI8 measured by masimo radical 7 equipment. | 1 minute after tidal volume challenge when tidal volume of patient is 8ml/kg
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of PVI8 measured by masimo radical 7 equipment. | 1 minute after tidal volume challenge, when tidal volume of patient is 8ml/kg.
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of Perfusion Index measured by masimo radical 7 equipment. | 1 minute before and 1 minte after tidal volume challenge (patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of Perfusion Index measured by masimo radical 7 equipment. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of Cardiac Index measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of Cardiac Index measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of Cardiac Output measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of Cardiac Output measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of Stroke Volume measured by electrical cardiometry and transoesophageal Doppler.. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of Stroke Volume measured by electrical cardiometry and transoesophageal Doppler.. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of Stroke Volume Index measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of Stroke Volume Index measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of Stroke Volume variation measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of Stroke Volume variation measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of Systemic vascular resistance measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of Systemic vascular resistance measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of Heart Rate measured by transoesophageal Doppler and masimo radical 7 equipment | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of Heart Rate measured by transoesophageal Doppler and masimo radical 7 equipment | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of central venous pressure measured by central venous catheter transducer. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of central venous pressure measured by central venous catheter transducer. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of Thoracic Fluid Content measured by electrical cardiometry. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of Thoracic Fluid Content measured by electrical cardiometry. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of corrected flow time measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of corrected flow time measured by electrical cardiometry and transoesophageal Doppler. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of contractility index measured by electrical cardiometry. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of contractility index measured by electrical cardiometry. | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of sensitivity of mean arterial blood pressure by invasive arterial blood pressure transducer | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves
Detection of specificity of mean arterial blood pressure by invasive arterial blood pressure transducer | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  By areas under the receiver operating characteristics (ROC) curves

OTHER OUTCOMES:
age | once when patient is recruited
  in years
sex | once when patient is recruited
  Male or female
Height | once when patient is recruited
  in meters
Actual body weight | once when patient is recruited
  in kilograms
Predicted body weight | once when patient is recruited
  in kilograms using equation for males = (50+2.3 ( height (inch)-60) while for females = ( 45.5 + 2.3 ( height (inch) -60)
BMI | once when patient is recruited
  kilograms/m2
comorbid diseases | once when patient is recruited
  names of diseases if present
operative time | immediately after the end of surgery
  in hours
measurement of compliance of the respiratory system from ventilator ml/cmH2O | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  ml/cmH2O
Measurement of plateau pressure from ventilator | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  cmH2O
Measurement of driving pressure in cmH2O | 1 minute before and 1 minute after tidal volume challenge (when patient's tidal volume 6 and 8 ml/kg)
  plateau pressure minus positive end expiratory pressure
preliminary suggestion of resected segment(s) of liver in hepatic resection operation | 10 minutes before beginning of operation
  number of segment(s)
Actual resected segment(s) of liver in hepatic resection operation | 5 minutes after completion of resection
  number of segment(s)

CONTACTS AND LOCATIONS:
Overall Officials: Magdy K Mohamed Khalil, M.D, Study Chair — National Liver Institute, Menoufia University; Mohamed F Mohamed El-Gayar, M.D, Study Director — Faculty of medicine, Fayoum University; Joseph M Botros, M.D, Study Director — Faculty of medicine, Fayoum University
Locations (1):
- National Liver Institute, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Results and Conclusion

REFERENCES:
- [Result] Tympa A, Theodoraki K, Tsaroucha A, Arkadopoulos N, Vassiliou I, Smyrniotis V. Anesthetic Considerations in Hepatectomies under Hepatic Vascular Control. HPB Surg. 2012;2012:720754. doi: 10.1155/2012/720754. Epub 2012 May 28. PMID 22690040
- [Result] Navarro LH, Bloomstone JA, Auler JO Jr, Cannesson M, Rocca GD, Gan TJ, Kinsky M, Magder S, Miller TE, Mythen M, Perel A, Reuter DA, Pinsky MR, Kramer GC. Perioperative fluid therapy: a statement from the international Fluid Optimization Group. Perioper Med (Lond). 2015 Apr 10;4:3. doi: 10.1186/s13741-015-0014-z. eCollection 2015. PMID 25897397
- [Result] Joshi GP. Intraoperative fluid restriction improves outcome after major elective gastrointestinal surgery. Anesth Analg. 2005 Aug;101(2):601-605. doi: 10.1213/01.ANE.0000159171.26521.31. PMID 16037184
- [Result] Smyrniotis V, Kostopanagiotou G, Theodoraki K, Tsantoulas D, Contis JC. The role of central venous pressure and type of vascular control in blood loss during major liver resections. Am J Surg. 2004 Mar;187(3):398-402. doi: 10.1016/j.amjsurg.2003.12.001. PMID 15006570
- [Result] Michard F, Teboul JL. Using heart-lung interactions to assess fluid responsiveness during mechanical ventilation. Crit Care. 2000;4(5):282-9. doi: 10.1186/cc710. Epub 2000 Sep 1. PMID 11094507
- [Result] Michard F, Schmidt U. Prediction of fluid responsiveness: searching for the Holy Grail. J Appl Physiol (1985). 2004 Aug;97(2):790-1; author reply 791. doi: 10.1152/japplphysiol.00021.2004. No abstract available. PMID 15247205
- [Result] Myatra SN, Prabu NR, Divatia JV, Monnet X, Kulkarni AP, Teboul JL. The Changes in Pulse Pressure Variation or Stroke Volume Variation After a "Tidal Volume Challenge" Reliably Predict Fluid Responsiveness During Low Tidal Volume Ventilation. Crit Care Med. 2017 Mar;45(3):415-421. doi: 10.1097/CCM.0000000000002183. PMID 27922879